CLINICAL TRIAL: NCT05254561
Title: Triple Intralesional Antigen Immunotherapy Versus Monoantigen in the Treatment of Multiple Recalcitrant Warts
Brief Title: Triple Antigen vs Monoantigen Immunotherapy for Warts
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Basma Magdy Elkholy, MD, Dr, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB# 6526/-15-11-2020
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Triple Intralesional Immunotherapy Combination in Multiple Recalcitrant Warts
Keywords: triple intralesional immunotherapy; Warts; tuberculin purified protein derivative; Candida antigen; Measles-Mumps-Rubella vaccine; combination immunotherapy
MeSH Terms: conditions — Warts | interventions — Tuberculin

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Investigator
Masking Description: Double masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- purified protein derivative (PPD) (Active Comparator): Group A
  Interventions: Biological: Intralesional antigen immunotherapy
- Candida antigen. (Active Comparator): Group B
  Interventions: Biological: Intralesional antigen immunotherapy
- Measles, Mumps and Rubella vaccine (MMR). (Active Comparator): Group C
  Interventions: Biological: Intralesional antigen immunotherapy
- Triple combination of PPD, Candida antigen and MMR (Active Comparator): Group D
  Interventions: Biological: Intralesional antigen immunotherapy

INTERVENTIONS:
Biological: Intralesional antigen immunotherapy — Randomized double-blinded comparative effectiveness and safety clinical trial
  Other Names: PPD, Candida antigen, and MMR

SUMMARY:
Warts can be resistant to treatment or return despite the use of many therapeutic modalities. Combining immunotherapy might contribute to better response rates, particularly in recalcitrant warts, which is a real therapeutic challenge. The purpose of this study was to assess the effectiveness and safety of a triple intralesional immunotherapy combination composed of PPD, Candida antigen and MMR versus either agent alone in the management of multiple recalcitrant warts.

DETAILED DESCRIPTION:
This study included 160 patients with multiple (>3 warts) recalcitrant (at least 6 months duration and who did not respond to at least 2 treatment modalities) warts of different sites, size and duration, with or without distant warts after approval of the Institutional Review Board of Faculty of medicine, Zagazig university. They were randomly assigned to one of four groups (each with 40 patients): PPD, Candida antigen, MMR, or combination of the 3 antigens. Injections into the biggest wart were repeated every two weeks until clearance or for a total of five sessions.

ELIGIBILITY:
Inclusion Criteria:

* Multiple (> 3 warts) recalcitrant (at least 6 months duration and who did not respond to at least 2 treatment modalities) warts of different sites, size and duration

Exclusion Criteria:

1. Patients with acute febrile illness or past history of asthma.
2. Allergic skin disorders such as generalized eczema and urticaria.
3. Past history of meningitis or convulsions.
4. Pregnancy or lactation.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Overall complete response of both treated and distant warts | within 12 weeks of starting treatment sessions (up to 1 month after the last session, maximum 5 sessions)
Immediate adverse effects | during and till 20 minutes after intralesional injection immunotherapy

SECONDARY OUTCOMES:
Distant wart clearance | within 12 weeks of starting sessions
Time to complete clearance | within 12 weeks of starting therapy
late adverse effects | after each session and till the end of sessions and 6 months-follow-up period
Recurrence | For 6 months after complete response

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig university, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Undecided